CLINICAL TRIAL: NCT02416258
Title: A Phase 2a Trial Evaluating the Anti-psoriatic Effect of LP0113 Aerosol Spray Compared With Its Vehicle and With Daivobet® Gel, LEO 90100 Aerosol Foam, Betamethasone Dipropionate Aerosol Spray and Calcipotriol Aerosol Spray in the Treatment of Psoriasis Vulgaris
Brief Title: A Psoriasis Plaque Test Trial With LP0113 Spray in Patients With Psoriasis Vulgaris (LP0113-1123)
Acronym: LP0113-1123
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: LP0113-1123; 2014-004759-30 (EudraCT Number)
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2017-05

CONDITIONS: Skin and Connective Tissue Diseases
Keywords: Psoriasis
MeSH Terms: conditions — Skin and Connective Tissue Diseases; Psoriasis | interventions — Aerosolized Particles and Droplets

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- LP0113 aerosol spray (Active Comparator): Calcipotriol (as monohydrate) 50 mcg/g and betamethasone (as dipropionate) 0.5 mg/g, topical
  Interventions: Drug: Aerosol spray vehicle; Drug: LEO 90100 aerosol foam; Drug: Betamethasone dipropionate aerosol spray; Drug: Calcipotriol aerosol spray; Drug: Daivobet® gel
- Aerosol spray vehicle (Placebo Comparator): No active ingredient, topical
  Interventions: Drug: LP0113 aerosol spray; Drug: LEO 90100 aerosol foam; Drug: Betamethasone dipropionate aerosol spray; Drug: Calcipotriol aerosol spray; Drug: Daivobet® gel
- LEO 90100 aerosol foam (Active Comparator): Calcipotriol (as monohydrate) 50 mcg/g and betamethasone (as dipropionate) 0.5 mg/g, topical
  Interventions: Drug: LP0113 aerosol spray; Drug: Aerosol spray vehicle; Drug: Betamethasone dipropionate aerosol spray; Drug: Calcipotriol aerosol spray; Drug: Daivobet® gel
- Betamethasone dipropionate aerosol spray (Active Comparator): Betamethasone (as dipropionate) 0.5 mg/g, topical
  Interventions: Drug: LP0113 aerosol spray; Drug: Aerosol spray vehicle; Drug: LEO 90100 aerosol foam; Drug: Calcipotriol aerosol spray; Drug: Daivobet® gel
- Calcipotriol aerosol spray (Active Comparator): Calcipotriol (as monohydrate) 50 mcg/g, topical
  Interventions: Drug: LP0113 aerosol spray; Drug: Aerosol spray vehicle; Drug: LEO 90100 aerosol foam; Drug: Betamethasone dipropionate aerosol spray; Drug: Daivobet® gel
- Daivobet® gel (Active Comparator): Calcipotriol (as monohydrate) 50 mcg/g and betamethasone (as dipropionate) 0.5 mg/g, topical
  Interventions: Drug: LP0113 aerosol spray; Drug: Aerosol spray vehicle; Drug: LEO 90100 aerosol foam; Drug: Betamethasone dipropionate aerosol spray; Drug: Calcipotriol aerosol spray

INTERVENTIONS:
Drug: LP0113 aerosol spray
  Arms: Aerosol spray vehicle; Betamethasone dipropionate aerosol spray; Calcipotriol aerosol spray; Daivobet® gel; LEO 90100 aerosol foam
Drug: Aerosol spray vehicle
  Arms: Betamethasone dipropionate aerosol spray; Calcipotriol aerosol spray; Daivobet® gel; LEO 90100 aerosol foam; LP0113 aerosol spray
Drug: LEO 90100 aerosol foam
  Arms: Aerosol spray vehicle; Betamethasone dipropionate aerosol spray; Calcipotriol aerosol spray; Daivobet® gel; LP0113 aerosol spray
Drug: Betamethasone dipropionate aerosol spray
  Arms: Aerosol spray vehicle; Calcipotriol aerosol spray; Daivobet® gel; LEO 90100 aerosol foam; LP0113 aerosol spray
Drug: Calcipotriol aerosol spray
  Arms: Aerosol spray vehicle; Betamethasone dipropionate aerosol spray; Daivobet® gel; LEO 90100 aerosol foam; LP0113 aerosol spray
Drug: Daivobet® gel
  Arms: Aerosol spray vehicle; Betamethasone dipropionate aerosol spray; Calcipotriol aerosol spray; LEO 90100 aerosol foam; LP0113 aerosol spray

SUMMARY:
The purpose of this study is to evaluate the anti-psoriatic effect of LP0113 aerosol spray compared to Daivobet® gel, LEO 90100 aerosol foam, betamethasone dipropionate in the aerosol spray vehicle, calcipotriol in the aerosol spray vehicle and aerosol spray vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent has been obtained
* Subjects with a diagnosis of psoriasis vulgaris with lesions located on arms, legs and/or trunk. The lesions must have a total size suitable for application of 6 different products.
* Age 18 years or above
* Outpatients
* Female subjects must be of either

  * non-childbearing potential, i.e. post-menopausal or have a confirmed clinical history of sterility (e.g. the subject is without a uterus or has tubal ligation) or,
  * child-bearing potential provided there is a confirmed negative pregnancy test prior to trial treatment to rule out pregnancy.

Exclusion Criteria:

* Female subjects who are breast feeding
* Systemic treatment with biological therapies, whether marketed or not, with a possible effect on psoriasis vulgaris within the following time periods prior to randomisation:

  * Etanercept - within 4 weeks prior to randomisation and during the trial
  * Adalimumab, infliximab - within 8 weeks prior to randomisation and during the trial
  * Ustekinumab - within 16 weeks prior to randomisation and during the trial
  * Other products - within 4 weeks/5 half-lives prior to randomisation and during the trial (whichever is longer)
* Systemic treatment with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, immunosuppressants) within the 4-week period prior to randomisation and during the trial,
* Subjects using phototherapy within the following time periods prior to randomisation and during the trial:

  * PUVA: 4 weeks
  * UVB: 2 weeks
* Subjects using one of the following topical drugs for the treatment of psoriasis within the 4 week period prior to randomisation and during the trial:

  * Potent or very potent (WHO group III-IV) corticosteroids
* Subjects using one of the following topical drugs for the treatment of psoriasis within 2 weeks prior to randomisation and during the trial:

  * WHO group I-II corticosteroids (except if used for treatment of scalp and/or facial psoriasis)
  * Topical retinoids, Vitamin D analogues, Topical immunomodulators (e.g. calcineurin inhibitors), Tar products, Salicylic acid
* Subjects using emollients on the selected plaques within 1 week before randomisation and during the trial
* Initiation of, or expected changes to concomitant medication that may affect psoriasis vulgaris (e.g., beta blockers, antimalarial drugs, lithium and ACE inhibitors) within 2 weeks prior to the randomisation and during the trial
* Subjects with current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Absolute change in Total Clinical Score (TCS) of clinical signs (sum of erythema, scaling and infiltration) | End of treatment compared to baseline - 4 weeks

SECONDARY OUTCOMES:
Absolute change in single clinical sign score: erythema, scaling, infiltration | End of treatment and individual visits compared to baseline - 4 weeks
Absolute Change in Total Clinical Score (TCS) | Individual visits compared to baseline - 4 weeks
Absolute change in total skin thickness and echo-poor band thickness | End of treatment compared to baseline - 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Pharmacologie Clinique Appliquée à la Dermatologie (CPCAD), Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en